CLINICAL TRIAL: NCT04560413
Title: Depression, Anxiety and SARS-CoV-2 Phobia in Post-stroke Patients During SARS-CoV-2 Pandemic
Brief Title: Depression, Anxiety and SARS-CoV-2 (Covid-19) Phobia in Post-stroke Patients
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSMEAH-KAEK 2020/41
Record Dates: First submitted 2020-09-20; First posted 2020-09-23 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV-2; Post-stroke Depression; Anxiety and Fear
Keywords: Anxiety; Post-stroke Depression; SARS-CoV-2; Phobia
MeSH Terms: conditions — Anxiety Disorders; Phobic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has begun, first in Wuhan, China, and then became a pandemic. The first SARS-CoV-2 case in Turkey was reported on March 11, 2020. People older than 65 years old became subject to lock down measures beginning on March 21, while people younger than 20 years old became subject to lock down measures beginning on April 03. A total lock down has been implemented a few times lasting between 3 to 4 days, especially at weekends. Several studies show that mental health problems could occur in public during the SARS-CoV-2 pandemic.

Depression and anxiety are a commonly known mental health issue in post-stroke patients. This patient population, who usually have to spend most of their time at home, remained completely at home and socially isolated due to the precautions required by the pandemic. Based on the above research evidence; depression, anxiety and phobia of SARS-CoV-2 may increase in the post stroke patients due to being in risk group and effects of measures taken against SARS-CoV-2 pandemic. Therefore, we aimed to assess the depression, anxiety and SARS-CoV-2 phobia in post stroke patients during SARS-CoV-2 outbreak, and to explore the potential influence factors.

DETAILED DESCRIPTION:
90 post-stroke patients who meet the working criteria were called by phone. All of them were followed up in the stroke outpatient clinic of the Physical Medicine and Rehabilitation Clinic. Only 77 patients were reached. Permission was asked for questioning from the patients reached. The health and social status of the patients who agreed to participate in the study during the SARS-CoV-2 pandemic period was questioned with the form we prepared. Form template included socio-demographic features, physical, and detailed medical histories. In addition, the fear based on the SARS-CoV-2 virus was examined with the Covid-19 phobia scale (CP19-S), while anxiety and depression were evaluated with the hospital anxiety and depression scale (HADS). Furthermore, Brunnstrom stages, Barthel index and functional ambulation classification (FAC), which was evaluated in the last 6 months, was recorded from the files to explore mobilization of the patients.

The C19P-S is a self-report instrument with a five-point Likert-type scale to assess the levels of SARS-CoV-2 phobia. All items are rated on a 5-point scale from "strongly disagree (1)" to "strongly agree (5)." The scores on the scale can range between 20 and 100 and a higher score indicates a greater phobia in the respected subscales and total scale. In the present study, total scale scores ranged from 20 to 100. The scale examines four main factors: psychological, psycho-somatic, economic and social HADS that includes anxiety and depression subscales. HADS is a self-report scale. It consists of 14 items, 7 of which are depression and 7 of which are symptoms of anxiety. Answers are evaluated in four Likert formats. The cutoff scores of the Turkish form of the HAD scale were determined as 10 for the anxiety subscale and 7 for the depression subscale. The purpose of the scale is not to make a diagnosis, but to determine the risk group by screening anxiety and depression in a short time in those with physical illness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old
* Post stroke patients
* Patients with mini mental state examination score above 24
* Patients who don't have aphasia
* Patients who were able to communicate in Turkish on the telephone

Exclusion Criteria:

* Patients under the 18 years old
* Patients who do not accept phone calls
* Patients with mini mental state examination score below 24
* Patients who have aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-stroke patients who aged over 18
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 3 months
  The Hospital Anxiety and Depression Scale evaluation includes a total of 14 questions (score range 0-3), which are scored to separately estimate anxiety and depressive status (7 questions each). The individual score for the anxiety and depression subscales may vary from 0 to 21. The aim of this scoring system is not to make an objective diagnosis, but to determine the current presence and tendency to anxiety or depression at the time of diagnosis. A HADS score of 8 to 10 is broadly accepted as indicating mild symptoms, a score between 11-16 suggests moderate anxiety or depression, and a score of 16 or more indicates severe anxiety or depressive symptoms
Covid 19 Phobia Scale | 3 months
  The Covid 19 Phobia Scale is a self-report instrument with a five-point Likert-type scale to assess the levels of SARS-CoV-2 phobia. All items are rated on a 5-point scale from "strongly disagree (1)" to "strongly agree (5)." The scores on the scale can range between 20 and 100 and a higher score indicates a greater phobia in the respected subscales and total scale. In the present study total scale scores ranged from 20 to 100. The scale examines four main factors: psychological, psycho-somatic, economic and social

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Silte Karamanlioglu, MD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital; Arzu Atici, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Gulcan Ozturk, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Pinar Akpinar, Assoc Prof, Study Director — Fatih Sultan Mehmet Training and Research Hospital; Feyza Unlu Ozkan, Assoc Prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Ilknur Aktas, Prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No